CLINICAL TRIAL: NCT03666442
Title: Early Evaluation of Chemosensitivity for Low-risk Stage II/III Rectal Cancer
Brief Title: Early Evaluation of Chemosensitivity for Low/Intermediated-risk Mid-low Stage II/III Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC-CT-2018
Record Dates: First submitted 2018-08-18; First posted 2018-09-11 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Rectal Cancer
Keywords: rectal cancer；; neoadjuvant Chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX

STUDY DESIGN:
Intervention Model Description: a group of patients receive 4 cycle of Xelox chemotherapy, MRI,TRUS, DE,endoscopy, blood DNA test,before, between and after chemotherapy was compared to detect the effect of chemotherapy in 2 cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemotherapy group (Experimental): patients receive 4 cycles of Xelox
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: XELOX — Xelox chemotherapy,that oxaliplatin 130mg/m2 d1,capecitabine 1000mg/m2 twice daily d1-14,every 3 weeks

SUMMARY:
Chemosensitivity of rectal cancer is not discussed clearly. With previous study, the investigators design this phase II trial to explore the effect of 2 cycles Xelox chemotherapy,so as to explore the early detection of sensitivity of tumor. With inclusion of early,intermediate,and bad stage II/III rectal cancer patients, four cycle of Xelox chemotherapy was given. After the second cycle, MRI,TRUS,DE,endoscopy,and blood DNA test was down to compare with these characteristics of four cycles.so that to detect the data about the chemosensitivity of tumor in the early stage.

DETAILED DESCRIPTION:
Chemosensitivity of rectal cancer is not discussed clearly. With previous study, the investigators design this phase II trial to explore the effect of 2 cycles Xelox chemotherapy,so as to explore the early detection of sensitivity of tumor. With inclusion of early,intermediate,and bad stage II/III rectal cancer patients, four cycle of Xelox chemotherapy was given. After the second cycle, MRI,TRUS,DE,endoscopy,and blood DNA test was down to compare with these characteristics of four cycles.so that to detect the data about the chemosensitivity of tumor in the early stage.In future, a phase III trial that explore the effect of radiation or surgery in these chemoresistant patients.

ELIGIBILITY:
Inclusion Criteria:

1. .endoscopy and biopsy verified rectal cancer within 12cm from anal verge;
2. .primary MRI, TRUS, abdomino-chest CT diagnosed early or intermediate or bad Stage II/III rectal cancer;
3. .age from 20-75;
4. .with informed consent;

Exclusion Criteria:

1. .refuse the further treatment after recruiting;
2. .diagnosis of peritoneal metastasis in the surgery;

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
tumor volume | At the end of Cycle 2 (each cycle is 3 weeks)
  tumor volume measured by MRI
tumor area in endoscopy | At the end of Cycle 2 (each cycle is 3 weeks)
  tumor area measured in endoscopy
tumor volume | At the end of Cycle 4 (each cycle is 3 weeks)
  tumor volume measured by MRI
tumor area in endoscopy | At the end of Cycle 4 (each cycle is 3 weeks)
  tumor area measured in endoscopy

SECONDARY OUTCOMES:
blood DNA test | At the end of Cycle 2 (each cycle is 3 weeks)
  blood DNA test
blood DNA test | At the end of Cycle 4 (each cycle is 3 weeks)
  blood DNA test
tumor thickness in TRUS | At the end of Cycle 4 (each cycle is 3 weeks)
  tumor thickness in TRUS
tumor thickness in TRUS | At the end of Cycle 2 (each cycle is 3 weeks)
  tumor thickness in TRUS

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, MD, Study Chair — West China Hospital
Locations (1):
- Guoxue Road 37#,West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schrag D, Weiser MR, Goodman KA, Gonen M, Hollywood E, Cercek A, Reidy-Lagunes DL, Gollub MJ, Shia J, Guillem JG, Temple LK, Paty PB, Saltz LB. Neoadjuvant chemotherapy without routine use of radiation therapy for patients with locally advanced rectal cancer: a pilot trial. J Clin Oncol. 2014 Feb 20;32(6):513-8. doi: 10.1200/JCO.2013.51.7904. Epub 2014 Jan 13. PMID 24419115
- [Result] Sclafani F, Cunningham D. Neoadjuvant chemotherapy without radiotherapy for locally advanced rectal cancer. Future Oncol. 2014 Nov;10(14):2243-57. doi: 10.2217/fon.14.127. PMID 25471037
- [Result] Birlik B, Obuz F, Elibol FD, Celik AO, Sokmen S, Terzi C, Sagol O, Sarioglu S, Gorken I, Oztop I. Diffusion-weighted MRI and MR- volumetry--in the evaluation of tumor response after preoperative chemoradiotherapy in patients with locally advanced rectal cancer. Magn Reson Imaging. 2015 Feb;33(2):201-12. doi: 10.1016/j.mri.2014.08.041. Epub 2014 Nov 13. PMID 25460330
- [Result] Zhang J, Cai Y, Hu H, Lan P, Wang L, Huang M, Kang L, Wu X, Wang H, Ling J, Xiao J, Wang J, Deng Y. Nomogram basing pre-treatment parameters predicting early response for locally advanced rectal cancer with neoadjuvant chemotherapy alone: a subgroup efficacy analysis of FOWARC study. Oncotarget. 2016 Jan 26;7(4):5053-62. doi: 10.18632/oncotarget.6469. PMID 26646794
- [Result] Koike J, Funahashi K, Yoshimatsu K, Yokomizo H, Kan H, Yamada T, Ishida H, Ishibashi K, Saida Y, Enomoto T, Katsumata K, Hisada M, Hasegawa H, Koda K, Ochiai T, Sakamoto K, Shiokawa H, Ogawa S, Itabashi M, Kameoka S. Efficacy and safety of neoadjuvant chemotherapy with oxaliplatin, 5-fluorouracil, and levofolinate for T3 or T4 stage II/III rectal cancer: the FACT trial. Cancer Chemother Pharmacol. 2017 Mar;79(3):519-525. doi: 10.1007/s00280-017-3243-7. Epub 2017 Feb 1. PMID 28150022
- [Result] Patel UB, Brown G, Machado I, Santos-Cores J, Pericay C, Ballesteros E, Salud A, Isabel-Gil M, Montagut C, Maurel J, Ramon-Ayuso J, Martin N, Estevan R, Fernandez-Martos C. MRI assessment and outcomes in patients receiving neoadjuvant chemotherapy only for primary rectal cancer: long-term results from the GEMCAD 0801 trial. Ann Oncol. 2017 Feb 1;28(2):344-353. doi: 10.1093/annonc/mdw616. PMID 28426108
- [Result] Chee CG, Kim YH, Lee KH, Lee YJ, Park JH, Lee HS, Ahn S, Kim B. CT texture analysis in patients with locally advanced rectal cancer treated with neoadjuvant chemoradiotherapy: A potential imaging biomarker for treatment response and prognosis. PLoS One. 2017 Aug 10;12(8):e0182883. doi: 10.1371/journal.pone.0182883. eCollection 2017. PMID 28797063
- [Result] Battersby NJ, How P, Moran B, Stelzner S, West NP, Branagan G, Strassburg J, Quirke P, Tekkis P, Pedersen BG, Gudgeon M, Heald B, Brown G; MERCURY II Study Group. Prospective Validation of a Low Rectal Cancer Magnetic Resonance Imaging Staging System and Development of a Local Recurrence Risk Stratification Model: The MERCURY II Study. Ann Surg. 2016 Apr;263(4):751-60. doi: 10.1097/SLA.0000000000001193. PMID 25822672
- [Result] Glynne-Jones R, Wyrwicz L, Tiret E, Brown G, Rodel C, Cervantes A, Arnold D; ESMO Guidelines Committee. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv22-iv40. doi: 10.1093/annonc/mdx224. No abstract available. PMID 28881920
- [Derived] Deng X, Wu Q, Bi L, Yu Y, Huang S, He D, Wu B, Gou H, Meng W, Qiu M, He Y, Wang Z. Early response to upfront neoadjuvant chemotherapy (CAPOX) alone in low- and intermediate-risk rectal cancer: a single-arm phase II trial. Br J Surg. 2021 Dec 17;109(1):121-128. doi: 10.1093/bjs/znab388. PMID 34792107
- See also: NCCN guideline — https://www.nccn.org/professionals/physician_gls/pdf/rectal.pdf